CLINICAL TRIAL: NCT01500395
Title: Hybrid Operation in Thoracic Aortic Dissection---Registry of China
Brief Title: Hybrid Operation in Thoracic Aortic Dissection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJ-20111126 -2
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Aorta Dissection; Aorta Aneurysm
Keywords: Aortic Diseases; Vascular Diseases; Cardiovascular Diseases; Treatment Outcome; Aorta Dissection; Aorta Aneurysm; Aorta pseudoaneurysm; Endovascular aortic repair; Hybrid operation; Debranching
MeSH Terms: conditions — Aortic Dissection; Aortic Aneurysm; Aortic Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stent Graft and open surgery: Hybrid Operations including debranching technique+Thoracic Endovascular Aortic Repair (TEVAR), Frozen elephant trunk technique, aortic arch replacement with concommitant TEVAR, et al.
  Interventions: Procedure: Hybrid operation

INTERVENTIONS:
Procedure: Hybrid operation — Hybrid Operations including debranching technique+Thoracic Endovascular Aortic Repair (TEVAR), Frozen elephant trunk technique, aortic arch replacement with concommitant TEVAR, et al. Devices include Medtronic Stent Graft（Medtronic Medtronic, Inc., US） Microport Stent Graft（Microport Co.,LTD.，Shanghai, China） Ankura Stent Graft（Lifetech Scientific Co.,LTD.，Shenzhen, China）.
  Other Names: Medtronic Stent Graft; Microport Stent Graft; Ankura Stent Graft

SUMMARY:
The purpose of this study is to investigate the short to mid term efficacy and safety of different hybrid operations who had complex aortic lesions, such as ascending aortic/arch aneurysm, pseudo-aneurysm, Stanford Type A dissection, retrograde Stanford Type B dissection, dissection with primary tear located in the aortic arch, et al.

DETAILED DESCRIPTION:
Aneurysms and dissection involving the ascending aorta and aortic arch have historically been treated with open surgical techniques, requiring cardiopulmonary bypass and deep hypothermic circulatory arrest (DHCA). Despite increasing experience and refinement of these procedures, there remains a substantial rate of morality and morbidity. The goal of hybrid operations is to re-construct the ascending aorta and aortic arch to cover the primary entry tear of the dissection and to remodel the aorta. Hybrid Operations including debranching technique+Thoracic Endovascular Aortic Repair (TEVAR), Frozen elephant trunk technique, aortic arch replacement with concommitant TEVAR, et al. The purpose of this study is to investigate the short to mid term efficacy and safety of different hybrid operations who had complex aortic lesions, such as ascending aortic/arch aneurysm, pseudo-aneurysm, Stanford Type A dissection, retrograde Stanford Type B dissection, dissection with primary tear located in the aortic arch, et al.

Primary outcome measure is all-cause mortality. Secondary outcome variables include conversion to stent and/or surgery, induced thrombosis of the false lumen, cardiovascular morbidity, aortic expansion (>5 mm/y of maximum diameter including true and false lumina), quality of life, and length of intensive care unit and hospital stay. The study designs to enroll 50 patients to be monitored for 24 months.

ELIGIBILITY:
Inclusion CriteriaInclusion Criteria:

* Ascending aortic/arch aneurysm
* Ascending aortic/arch pseudo-aneurysm
* Stanford Type A dissection
* Retrograde Stanford Type B dissection
* Unclassified dissection with primary tear located in the aortic arch
* Able to tolerate endotracheal intubation and general anesthesia
* Subject's anatomy must meet the anatomical criteria to receive that implanted device
* The subject or legal guardian understands the nature of the study and agrees to its provisions on a written informed consent form
* Availability for the appropriate follow-up visits during the follow-up period
* Capability to follow all study requirements

Exclusion Criteria:

* ASA classification = V
* Severe renal insufficiency defined as SVS risk renal status = 3
* Severe respiratory insufficiency defined as SVS risk pulmonary status = 3
* Presence of connective tissue disease
* Active infection or active vasculitides
* Pregnant woman or positive pregnancy test
* Myocardial infarction or cerebrovascular accident within 6 weeks prior to study enrollment
* Subject has had a cerebral vascular accident (CVA) within 2 months.
* History of drug abuse
* Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
* Subject has a known allergy or intolerance to the device components.
* Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.
* Subject has a co-morbidity causing expected survival to be less than 1 year.
* Enrolment in another clinical study
* Unwillingness to cooperate with study procedures or follow-up visits

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Thoracic Aortic Dissection
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative MACE | 12 months
  Cumulative MACE (including death, rupture, paraplegia, aneurysm formation et al)

SECONDARY OUTCOMES:
Endoleak | 12 months
  Endoleak of all types from the stent graft
Stent-graft migration/kinking | 12 months
  Stent-graft migration, stenosis, kinking and other conditions requiring re-intervention
Cumulative cerebrovascular events | 12 months
  Cumulative cerebrovascular events as bleeding, thrombosis, paraplegia, transient unconsciousness, et al.
Liver/Kidney dysfunction | 12 months
  Liver dysfunction including jaundice，transaminase elevation 1.5 times more than normal, et al.
  Kidney dysfunction including oliguria, anuria, Creatinine/BUN elevation 1.5 times more than normal, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Dinghua Yi, M.D., Ph.D, Principal Investigator — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University; Jian Yang, M.D., Ph.D., Study Director — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University; Weixun Duan, M.D., Ph.D., Study Director — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University; Shiqiang Yu, M.D., Study Director — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University; Jincheng Liu, M.D., Study Director — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University; Wensheng Chen, M.D., Study Director — Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Cardiovascular Surgery of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China